CLINICAL TRIAL: NCT06814535
Title: A Comparative Study on the Impact of Trigger Points Injection of Platelet Rich Plasma Versus Botulinum Toxin a on the Relief of Jaw Muscles Myofascial Pain
Brief Title: A Comparative Study on the Impact of Trigger Points Injection of Platelet Rich Plasma Versus Botulinum Toxin on the Relief of Jaw Muscles Myofascial Pain
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, asmaa abdelrahman abdelhakeem sayed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD_CU_9122023
Record Dates: First submitted 2025-01-26; First posted 2025-02-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Patients with Jaw Muscles Myofascial Pain
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (3):
- Botulinum toxin A (Active Comparator): 20 Patients with Myofascial pain will be injected by 5 units botulinum toxin A per trigger point in masseter and/or temporalis
  Interventions: Drug: Botulinum Toxin A / Botulinum Toxin A
- Platelet rich plasma (Active Comparator): 20 patients with Myofascial pain will be injected by .5 ml PRP solution per trigger point in masseter and/or temporalis
- Physiologic saline (Placebo Comparator): 20 patients with Myofascial pain will be injected by.5 ml physiologic saline per each trigger point

INTERVENTIONS:
Drug: Botulinum Toxin A / Botulinum Toxin A — Botulinum toxin type A
  Arms: Botulinum toxin A
Drug: Platelet rich plasma — Plasma that contains concentrated platelets
Drug: Saline -- placebo comparator — Physiological saline .9 %

SUMMARY:
This study aims at comparing the effect of trigger points injection of platelet rich plasma and botulinum toxin a on the relief of jaw muscles Myofascial pain .

The 1st group includes 20 patients who are supposed to receive 5 units of botulinum toxin A per trigger point in masseter and/or temporalis muscles.

The 2nd group will receive ,5 ml of PRP per trigger point in masseter and/or temporalis muscles.

The 3rd group will receive .5 ml of physiologic saline per each trigger point in masseter and/or temporalis muscles.

The 1st follow up session will be after 1 week then 1 month then 3 months . The patients are advised to limit excessive Mouth opening, yawning or singing. And when pain episode , theta re advised to take only paracetamol as analgesic drug .

At the follow up sessions ، measuring the interincisal opening , pressure pain threshold using algometer , VAS to measure the intensity of pain , Likert scale , current pain intensity, worst pain intensity and the need to take analgesics in Numbers.

Then comparing the results of these groups to end in rejecting the null hypothesis which says there's an equivalence between the 3 types of injected solutions or accepting it .

ELIGIBILITY:
Inclusion Criteria:

* patient with myofascial trigger points in masseter or temporalis previously ----*identified by manual palpation.

  * 18 years or More "Willingness to follow instructions.

Exclusion Criteria:

* therapeutic intervention for myofascial pain in the last view months such as taking medications for pain control or wearing an occlusal splint.

  * Clinical conditions as pregnancy
  * Medical problems that will interfere with the procedure as bleeding disorders.
  * Cognitive impairment or present inadequate cooperation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold | 3 months
  The amount of force per kilogram needed to induce pain in patients with myofascial pain at the trigger point..
  Will be measured using the algometer which presses on the trigger point to induce pain by force measured in kilograms/cm2 If the reading increased among the treatment visits , this means better outcome and decreased pain intensity with effectiveness of the treatment
Current pain intensity | 3 months
  The amount of pain on VAS at the time of examination from 0-10 With 0 no pain which increases to reach 10 ( the highest pain intensity).. Decrease in pain intensity means better outcome
Worst pain intensity | 3 months
  The worst pain the patient had suffered from on the previous duration. Using visual analogue scale from (0-10) with 0 least pain and 10 worst pain .
  Decrease in pain intensity means better outcome

SECONDARY OUTCOMES:
Inter incisal opening | 3 months
  The measurement in millimeters of the distance between the incisal edge of the upper incisor and the lower incisor Using calibers to measure the effect of myofascial pain on decreasing muscle spasm and the effectiveness of the treatment by time.
  Increased degree of mouth opening meaning the muscles had relaxed and trigger points released
Patient satisfaction | 3 months
  Will be measured by Likert scale by faces to indicate whether the treatment was satisfactory to the patient or not and to which degree .it affected their quality of life
The need for analgesics | 3 months
  The patient will count how many Paracetamol tabs he took at the time from the last visit till now.
  With decreased amount of analgesics taken between the visits means better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided